CLINICAL TRIAL: NCT05215249
Title: Transnasal Humidified High-Flow Oxygen Delivery (Optiflow) vs. Conventional Tubeless Anesthesia for the Prevention of Desaturations During Pediatric Laryngeal Papilloma Removal
Brief Title: Optiflow vs. Convential Anesthesia During Pediatric Laryngeal Papilloma Removal
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB approval not received
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Nita Sahani, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019P001552
Record Dates: First submitted 2020-02-21; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Laryngeal Papilloma, Recurrent
MeSH Terms: conditions — Recurrent respiratory papillomatosis

STUDY DESIGN:
Intervention Model Description: randomized crossover study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Patient will receive conventional tubeless anesthesia
- High Flow Oxygen Delivery (Experimental): Patient will receive Transnasal humidified high-flow oxygen delivery (Optiflow)
  Interventions: Procedure: Transnasal humidified high-flow oxygen delivery

INTERVENTIONS:
Procedure: Transnasal humidified high-flow oxygen delivery — The Optiflow system consists of an apparatus that is capable of delivering humidified oxygen, room air, or a mixture of variable oxygen concentration. The oxygen concentration can be precisely varied from 21-100% (or 0.21 - 1.00 FiO2). The gas is warmed to 37°C with a 100% relative humidity. The humidified and warmed gas can be delivered to the patient at high-flows (up to 70 L/min) using various delivery mechanisms. The investigators will be using a nasal cannula to deliver high flow oxygen (2-3 L/kg/min) to the patient.
  Other Names: Optiflow
  Arms: High Flow Oxygen Delivery

SUMMARY:
This is a randomized cross over study of high flow oxygen delivery via nasal cannula vs. conventional tubeless anesthesia for patients undergoing dubulking surgery for laryngeal papilloma. Ten patients aged 2-17 with laryngeal papilloma that are eligible for debulking surgery will be consented and enrolled.

DETAILED DESCRIPTION:
This trial will be a randomized unmasked open-label study of Transnasal humidified high-flow oxygen/air delivery compared to conventional tubeless anesthesia during airway surgery in pediatric patients. This will be a single center study at MEE main campus on 243 Charles St, Boston, MA for the use of the high-flow oxygen delivery device.

Two study arms will be used in this study. Subjects will be treated with both study arms over the course of two study visits. Enrolled patients will be patients that present themselves routinely for removal of laryngeal papilloma. These patients, once enrolled, will be randomized to either receive conventional tubeless anesthesia or standard anesthesia with the addition of transnasal high-flow oxygen/air for their next scheduled anesthetic. Oxygen flows for the high-flow nasal cannula will be titrated down to achieve a FiO2 value of 21% during lasering. The anesthesia method not chosen will be used for the following anesthetic for each patient. Intraoperatively patients will be monitored for number of desaturations below 90 percent, length of these desaturations and severity, number and type of interventions necessary by the anesthesiologist, and number of intubations necessary by the anesthesiologist. Flow rates appropriate for the age of the patient will be used and also be recorded within these cases. Adverse events and complications will also be recorded for both anesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of laryngeal papilloma via endoscopic exam by a pediatric ENT surgeon. And the expectation that he or she will require multiple debulking surgeries.
2. Age 2-17 years old at time of consent and both surgeries.
3. Parent/guardian consent and patient assent has been given.

Exclusion Criteria:

1. Patients with nasal obstructions or are otherwise not candidates for high flow oxygen delivery via nasal cannula.
2. Patients with underlying complicating pulmonary diseases like severe asthma, pulmonary hypertension, or ongoing pneumonia.
3. Pregnant patients.
4. Absence of parent or legal guardian able to provide written consent.
5. Patients who in the opinion of the investigator would not be good candidates for debulking surgery.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | End of study
  The primary objective of this study is to investigate the effects of transnasal humidified high-flow oxygen/air system to maintain safe intraoperative oxygen saturations in pediatric patients undergoing procedures for removal of laryngeal papilloma, thereby improving the quality of care. Number, duration and severity of intraoperative desaturations below 90 percent.